CLINICAL TRIAL: NCT00294086
Title: A 12-Week Multicenter, 2-Arm Regimen, Exploratory Study to Evaluate the Tolerability and Safety of Valsartan Administered Once Daily vs Daily, in Patients With Stable, Chronic Heart Failure (NYHA Class Ll-lll)
Brief Title: A Study of Valsartan Administered Once Daily Versus Twice Daily, in Patients With Stable, Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Study Director, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489BUS70
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Heart Failure
Keywords: valsartan,; chronic heart failure,
MeSH Terms: interventions — Valsartan; BID protein, human

INTERVENTIONS:
Drug: valsartan 160 mg
Drug: valsartan 160 mg BID

SUMMARY:
This study will evaluate the tolerability and safety of valsartan in patients with stable, chronic heart failure (NYHA Class ll-lll). The 12-week double blind study has a 2-week (maximum) screening, and a 10-week active treatment phase. In each of the treatment arms (QD and BID), patients are up-titrated to a maximum valsartan total daily dose of 320 mg. Patients remain on their prior CHF standard care therapy throughout the study period, and the up-titration of valsartan is based on patient tolerability.

ELIGIBILITY:
Inclusion Criteria

* Males or females aged 18 years or older
* Diagnosis of chronic heart failure (CHF), in NYHA Class ll-lll beginning at least 3 months prior to Visit 1
* Patients must remain on their prior standard care CHF therapy

Exclusion Criteria

* Diagnosis of severe hypertension (SBP>180 and DBP>110 mm Hg)
* Right heart failure due to pulmonary disease
* Presence of rapidly deteriorating heart failure
* MI or cardiac surgery, including PTCA within 3 months of Visit 1
* Unstable angina or coronary artery disease likely to require CABG or PTCA
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Tolerability as assessed by laboratory tests for potassium, creatinine, and on systolic blood pressure, symptoms of low blood pressure, and symptoms of heart failure

SECONDARY OUTCOMES:
Patients reaching target dose at 10 weeks
Change from baseline in systolic blood pressure at each study visit
Change from baseline in diastolic blood pressure at each study visit
Change from baseline in blood potassium at each study visit
Change from baseline in blood creatinine at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Anand IS, Deswal A, Kereiakes DJ, Purkayastha D, Zappe DH. Comparison of once-daily versus twice-daily dosing of valsartan in patients with chronic stable heart failure. Vasc Health Risk Manag. 2010 Aug 9;6:449-55. PMID 20730060